CLINICAL TRIAL: NCT05185349
Title: Experiences and Perceived Needs Among Parents of Children Exposed to Potentially Traumatic Events: a Qualitative Inquiry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0700
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress; Child and Adolescent Psychiatry; Parental perceived needs
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at exploring qualitatively experiences and perceived needs among parents of children exposed to potentially traumatic events, including their attitudes and understanding of trauma and resilience, their perceptions of their parental role in the peri-traumatic period, and their expectations of a family intervention for post-traumatic stress. This will ultimately guide future research to develop and design and intervention that would be tailored to their needs and expectations

ELIGIBILITY:
Inclusion criteria:

* Being a parent of a child aged 7-17
* exposed or who recently revealed a potentially traumatic event in the past six months

Exclusion criteria: Abusive parent Child and/or parent with intellectual deficiency

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study aims at exploring experiences and perceived needs among parents of children recently exposed (or who recently revealed) a potentially traumatic event.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Experiences and attitudes around trauma | 1 day
  Qualitative inquiry into parents' experiences in the post-traumatic period of their child

SECONDARY OUTCOMES:
Perceptions of parental role and ways to cope | 1 day
  Qualitative inquiry into parental's Perceptions of parental role and ways to cope

CONTACTS AND LOCATIONS:
Overall Officials: Diane Purper-Ouakil, M.D., Ph. D., Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC